CLINICAL TRIAL: NCT00640042
Title: AVINZA Control of Chronic Pain, Effectiveness and Safety Study (ACCESS 2008) A Multi-Center Study to Evaluate the Effectiveness and Tolerability of AVINZA for Chronic Moderate-Severe Pain: A Focus on Risk Minimization Assessment, Intervention and Outcomes
Brief Title: Evaluation of Risk Minimization, Assessment and Outcomes in Patients With Chronic Pain Taking Avinza
Acronym: ACCESS 2008
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K284-07-4001
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Pain
Keywords: pain; opioid; abuse; moderate-severe pain requiring continuous, around-the-clock opioid therapy for an extended period of time
MeSH Terms: conditions — Pain | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: morphine sulfate extended release capsules

INTERVENTIONS:
Drug: morphine sulfate extended release capsules — 30 mg, 60 mg, 90 mg, 120 mg morphine will be prescribed by the Investigator in accordance with the AVINZA prescribing information.
  Other Names: AVINZA

SUMMARY:
The purpose of this study is to provide information in a broad, "real world" population of chronic pain patients assessing both pain control with AVINZA as well as the potential risk for misuse and abuse.

DETAILED DESCRIPTION:
Pain affects more Americans than diabetes, heart disease and cancer combined and although it is one of the earliest known ailments, pain is still without a universal cure. It is estimated that only about 25% of patients with chronic pain receive adequate analgesia.

Long-term treatment of chronic pain with opioids is recognized as an important treatment option for patients with moderate-severe pain related to cancer and other chronic serious illnesses. AVINZA (morphine sulfate extended-release capsules) was approved for marketing by the Food and Drug Administration (FDA) in 2002 as a once daily treatment for the relief of moderate to severe pain requiring continuous opioid therapy for an extended period of time. While opioids, such as AVINZA, are beneficial in the management of chronic pain, they are sometimes associated with illicit activities. Misuse, abuse and diversion of controlled prescription drugs, particularly opioids, are problems that have increased dramatically in the United States (U.S.) since the 1990s.

This study will follow the Federation of State Medical Boards Model Policy for the Use of Controlled Substances for the Treatment of Pain. Patients will be counseled on the proper storage and destruction of unused AVINZA in accordance with federal and applicable state laws. A universal precautions approach to chronic pain management (KAIR) will be utilized in this study. Although not validated as a risk assessment and management instrument, KAIR is designed to assist clinicians with responsibly managing chronic moderate-severe pain patients prescribed AVINZA. The KAIR tools will be used by the Investigator to determine the level of monitoring required based on the patient's potential risk for opioid misuse or abuse (KAIR level). Investigators and staff participating in this study will be required to participate in a training program on the counseling to be given, procedures to be followed and tools to be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an adult (greater than or equal to 21 years old
* Patient has chronic (greater than or equal to 3 months) moderate-severe pain who, at the discretion of the Investigator, requires an around-the-clock opioid for optimal analgesia. Patients may be opioid naïve (not currently on an opioid) or opioid tolerant. Opioid naïve patients with a pain score of greater than or equal to 4 on an 11-point NRS (numerical rating scale. OR Opioid tolerant patients experiencing suboptimal response (i.e. pain score of greater than or equal to 4) or unacceptable side effects to sustained release opioids or short-acting opioids.
* Patient is able to read and understand English and comply with protocol requirements.

Exclusion Criteria:

A patient who meets ANY of the following exclusion criteria will not be enrolled:

* Hypersensitivity to morphine, morphine salts, or any components of AVINZA
* Respiratory depression (slowed breathing)
* Acute or severe bronchial asthma or severe chronic obstructive pulmonary disease (COPD)
* Currently has or is suspected of having paralytic ileus
* Requires a daily dose of AVINZA greater than 1600mg/day
* Patient is abusing alcohol
* Pregnancy or breast feeding
* Currently taking AVINZA
* Patient unwilling to sign the Treatment Agreement
* Life expectancy is less than 2 months
* Migraine as the primary pain score
* Patient resides in a hospital or nursing home
* Patient has had more than 2 surgeries for low back pain
* Patient is anticipated to require major surgery or steroid injections for chronic pain over the next 12 weeks

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1570 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Siegel, MD, Study Director — King Pharmaceuticals is now a wholly owned subsidiary of Pfizer
Locations (323):
- United States (317):
  - Adamsville, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sun City, Arizona
  - Sun Lakes, Arizona
  - Tucson, Arizona
  - Burlingame, California
  - Castro Valley, California
  - Fountain Valley, California
  - Hemet, California
  - Lakewood, California
  - Livermore, California
  - Los Gatos, California
  - Murrieta, California
  - Nevada City, California
  - Oakland, California
  - Rocklin, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - West Hollywood, California
  - Whittier, California
  - Yuba City, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Fort Collins, Colorado
  - Northglenn, Colorado
  - Thornton, Colorado
  - Wheat Ridge, Colorado
  - Manchester, Connecticut
  - Milford, Connecticut
  - New Haven, Connecticut
  - North Haven, Connecticut
  - Norwich, Connecticut
  - Georgetown, Delaware
  - Milton, Delaware
  - Wilmington, Delaware
  - Apopka, Florida
  - Bradenton, Florida
  - Brandon, Florida
  - Cape Coral, Florida
  - Daytona Beach, Florida
  - DeLand, Florida
  - Delray Beach, Florida
  - Deltona, Florida
  - Dunnellon, Florida
  - Estero, Florida
  - Eustis, Florida
  - Loxahatchee Groves, Florida
  - Maitland, Florida
  - Margate, Florida
  - Miami, Florida
  - Mt. Dora, Florida
  - New Smyrna Beach, Florida
  - North Miami Beach, Florida
  - Oakland Park, Florida
  - Oldsmar, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Oviedo, Florida
  - Pembroke Pines, Florida
  - Port Richey, Florida
  - Royal Palm Beach, Florida
  - South Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Augusta, Georgia
  - Cave Spring, Georgia
  - Conyers, Georgia
  - Covington, Georgia
  - Decatur, Georgia
  - Rome, Georgia
  - Statesboro, Georgia
  - Sugar Hill, Georgia
  - Rexburg, Idaho
  - Clinton, Illinois
  - Crestwood, Illinois
  - Creve Coeur, Illinois
  - Danville, Illinois
  - DeKalb, Illinois
  - Elmwood Park, Illinois
  - Flossmoor, Illinois
  - Gurnee, Illinois
  - Lockport, Illinois
  - Maryville, Illinois
  - Morton, Illinois
  - Naperville, Illinois
  - Oak Park, Illinois
  - Pekin, Illinois
  - Peoria, Illinois
  - St. Charles, Illinois
  - Washington, Illinois
  - Zion, Illinois
  - Anderson, Indiana
  - Evansville, Indiana
  - Franklin, Indiana
  - Highland, Indiana
  - Indianapolis, Indiana
  - La Porte, Indiana
  - Lawrenceburg, Indiana
  - Newburgh, Indiana
  - Rushville, Indiana
  - Seymour, Indiana
  - Whiteland, Indiana
  - Des Moines, Iowa
  - Le Claire, Iowa
  - Newton, Iowa
  - Kansas City, Kansas
  - Lansing, Kansas
  - Shawnee, Kansas
  - Florence, Kentucky
  - London, Kentucky
  - Louisville, Kentucky
  - Monticello, Kentucky
  - Russell Springs, Kentucky
  - Somerset, Kentucky
  - Baltimore, Maryland
  - Chester, Maryland
  - Havre de Grace, Maryland
  - Ocean City, Maryland
  - Brockton, Massachusetts
  - Springfield, Massachusetts
  - Bloomfield Hills, Michigan
  - Clarkston, Michigan
  - Clinton, Michigan
  - Dearborn, Michigan
  - Dearborn Heights, Michigan
  - Farmington Hills, Michigan
  - Grand Rapids, Michigan
  - Lansing, Michigan
  - Leslie, Michigan
  - Livonia, Michigan
  - Mason, Michigan
  - Muskegon, Michigan
  - Northville, Michigan
  - Okemos, Michigan
  - Owosso, Michigan
  - Pigeon, Michigan
  - Rochester Hills, Michigan
  - Southgate, Michigan
  - Sterling Heights, Michigan
  - Troy, Michigan
  - Waterford, Michigan
  - Cold Spring, Minnesota
  - Ballwin, Missouri
  - Cape Girardeau, Missouri
  - Chesterfield, Missouri
  - Clinton, Missouri
  - Florissant, Missouri
  - Hazelwood, Missouri
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - Mexico, Missouri
  - Mount Vernon, Missouri
  - Platte City, Missouri
  - Raymore, Missouri
  - Saint Charles, Missouri
  - Saint Joseph, Missouri
  - St Louis, Missouri
  - Warrenton, Missouri
  - Washington, Missouri
  - Weston, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Atco, New Jersey
  - Blackwood, New Jersey
  - Bloomfield, New Jersey
  - Brigantine, New Jersey
  - East Orange, New Jersey
  - Green Brook, New Jersey
  - Irvington, New Jersey
  - Iselin, New Jersey
  - Jersey City, New Jersey
  - Kenilworth, New Jersey
  - Lakewood, New Jersey
  - Mays Landing, New Jersey
  - Millburn, New Jersey
  - Nutley, New Jersey
  - Scotch Plains, New Jersey
  - South Bound Brook, New Jersey
  - Totowa, New Jersey
  - Union, New Jersey
  - Wenonah, New Jersey
  - Westville, New Jersey
  - Brooklyn, New York
  - Glendale, New York
  - Kenmore, New York
  - Mayville, New York
  - New York, New York
  - Orchard Park, New York
  - Port Jefferson Station, New York
  - Rochester, New York
  - Staten Island, New York
  - Suffern, New York
  - Asheboro, North Carolina
  - Jacksonville, North Carolina
  - Raleigh, North Carolina
  - Akron, Ohio
  - Ashtabula, Ohio
  - Bowling Green, Ohio
  - Canal Winchester, Ohio
  - Cincinnati, Ohio
  - Cuyahoga Falls, Ohio
  - Dayton, Ohio
  - Defiance, Ohio
  - Fairfield, Ohio
  - Fremont, Ohio
  - Gahanna, Ohio
  - Genoa, Ohio
  - Hamilton, Ohio
  - Kent, Ohio
  - Kingston, Ohio
  - Lancaster, Ohio
  - Maumee, Ohio
  - New Lexington, Ohio
  - Perrysburg, Ohio
  - Pickerington, Ohio
  - Springboro, Ohio
  - Stow, Ohio
  - Toledo, Ohio
  - Warren, Ohio
  - Youngstown, Ohio
  - Stillwater, Oklahoma
  - Estacada, Oregon
  - Eugene, Oregon
  - Lake Oswego, Oregon
  - Milwaukie, Oregon
  - Oregon City, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Tualatin, Oregon
  - Aliquippa, Pennsylvania
  - Archbald, Pennsylvania
  - Aston Mills, Pennsylvania
  - Avoca, Pennsylvania
  - Bala-Cynwyd, Pennsylvania
  - Bensalem, Pennsylvania
  - Carbondale, Pennsylvania
  - Chicora, Pennsylvania
  - Clarks Summit, Pennsylvania
  - Collegeville, Pennsylvania
  - Conneaut Lake, Pennsylvania
  - Cowansville, Pennsylvania
  - Downingtown, Pennsylvania
  - Doylestown, Pennsylvania
  - Drexel Hill, Pennsylvania
  - Drums, Pennsylvania
  - Dublin, Pennsylvania
  - Elizabeth, Pennsylvania
  - Elkins Park, Pennsylvania
  - Ford City, Pennsylvania
  - Greensburg, Pennsylvania
  - Honesdale, Pennsylvania
  - King of Prussia, Pennsylvania
  - Levittown, Pennsylvania
  - McKeesport, Pennsylvania
  - Montrose, Pennsylvania
  - Moon Township, Pennsylvania
  - Morrisville, Pennsylvania
  - Mount Pleasant, Pennsylvania
  - New Castle, Pennsylvania
  - New Wilmington, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Phoenixville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Royersford, Pennsylvania
  - Scranton, Pennsylvania
  - Shippensburg, Pennsylvania
  - Southampton, Pennsylvania
  - Springfield, Pennsylvania
  - Stoneboro, Pennsylvania
  - Union City, Pennsylvania
  - Warminster, Pennsylvania
  - Wilkes-Barre, Pennsylvania
  - Yardley, Pennsylvania
  - Camden, South Carolina
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Greer, South Carolina
  - Marion, South Carolina
  - West Columbia, South Carolina
  - Ashland City, Tennessee
  - Collierville, Tennessee
  - Dyersburg, Tennessee
  - Hendersonville, Tennessee
  - Hermitage, Tennessee
  - Lebanon, Tennessee
  - McKenzie, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Newport, Tennessee
  - Springfield, Tennessee
  - Sweetwater, Tennessee
  - Woodbury, Tennessee
  - Arlington, Texas
  - Fort Worth, Texas
  - Irving, Texas
  - Rusk, Texas
  - Southlake, Texas
  - Layton, Utah
  - South Jordan, Utah
  - West Jordan, Utah
  - West Valley City, Utah
  - Annandale, Virginia
  - Ashburn, Virginia
  - Fairfax, Virginia
  - Falls Church, Virginia
  - Lynchburg, Virginia
  - Reston, Virginia
  - Edmonds, Washington
  - Marysville, Washington
  - Olympia, Washington
  - Seattle, Washington
  - Huntington, West Virginia
  - Milwaukee, Wisconsin
- Puerto Rico (6):
  - Carolina
  - Cidra
  - Hato Rey
  - Juncos
  - Ponce
  - San Juan

REFERENCES:
- [Background] The American Pain Foundation. Pain Facts & Figures. January 2007. Available from http://www.painfoundation.org/print.asp?file=Newsroom/PainFacts.htm.
- [Background] Weiner KA. The decade of pain control and research. The Pain Practitioner. 2003 Spring;13(1):3-4.
- [Background] Joranson DE, Berger JW. Regulatory issues in pain management. J Am Pharm Assoc (Wash). 2000 Sep-Oct;40(5 Suppl 1):S60-1. PMID 11029873
- [Background] Caldwell JR, Rapoport RJ, Davis JC, Offenberg HL, Marker HW, Roth SH, Yuan W, Eliot L, Babul N, Lynch PM. Efficacy and safety of a once-daily morphine formulation in chronic, moderate-to-severe osteoarthritis pain: results from a randomized, placebo-controlled, double-blind trial and an open-label extension trial. J Pain Symptom Manage. 2002 Apr;23(4):278-91. doi: 10.1016/s0885-3924(02)00383-4. PMID 11997197
- [Background] Rauck RL, Bookbinder SA, Bunker TR, Alftine CD, Ghalie R, Negro-Vilar A, de Jong E, Gershon S. The ACTION study: a randomized, open-label, multicenter trial comparing once-a-day extended-release morphine sulfate capsules (AVINZA) to twice-a-day controlled-release oxycodone hydrochloride tablets (OxyContin) for the treatment of chronic, moderate to severe low back pain. J Opioid Manag. 2006 May-Jun;2(3):155-66. doi: 10.5055/jom.2006.0025. PMID 17319449
- [Background] Rauck RL, Bookbinder SA, Bunker TR, Alftine CD, Ghalie R, Negro-Vilar A, de Jong E, Gershon S. A randomized, open-label study of once-a-day AVINZA (morphine sulfate extended-release capsules) versus twice-a-day OxyContin (oxycodone hydrochloride controlled-release tablets) for chronic low back pain: the extension phase of the ACTION trial. J Opioid Manag. 2006 Nov-Dec;2(6):325-8, 331-3. doi: 10.5055/jom.2006.0048. PMID 17326594
- [Background] Rosenthal M, Moore P, Groves E, Iwan T, Schlosser LG, Dziewanowska Z, Negro-Vilar A. Sleep improves when patients with chronic OA pain are managed with morning dosing of once a day extended-release morphine sulfate (AVINZA): findings from a pilot study. J Opioid Manag. 2007 May-Jun;3(3):145-54. doi: 10.5055/jom.2007.0052. PMID 18027540
- [Background] Katz NP, Adams EH, Chilcoat H, Colucci RD, Comer SD, Goliber P, Grudzinskas C, Jasinski D, Lande SD, Passik SD, Schnoll SH, Sellers E, Travers D, Weiss R. Challenges in the development of prescription opioid abuse-deterrent formulations. Clin J Pain. 2007 Oct;23(8):648-60. doi: 10.1097/AJP.0b013e318125c5e8. PMID 17885342
- [Background] Ives TJ, Chelminski PR, Hammett-Stabler CA, Malone RM, Perhac JS, Potisek NM, Shilliday BB, DeWalt DA, Pignone MP. Predictors of opioid misuse in patients with chronic pain: a prospective cohort study. BMC Health Serv Res. 2006 Apr 4;6:46. doi: 10.1186/1472-6963-6-46. PMID 16595013
- [Background] Gourlay DL, Heit HA, Almahrezi A. Universal precautions in pain medicine: a rational approach to the treatment of chronic pain. Pain Med. 2005 Mar-Apr;6(2):107-12. doi: 10.1111/j.1526-4637.2005.05031.x. PMID 15773874
- [Derived] Setnik B, Roland CL, Pixton GC, Sommerville KW. Prescription opioid abuse and misuse: gap between primary-care investigator assessment and actual extent of these behaviors among patients with chronic pain. Postgrad Med. 2017 Jan;129(1):5-11. doi: 10.1080/00325481.2017.1245585. Epub 2016 Oct 26. PMID 27782769

RESULTS

PARTICIPANT FLOW:
Groups:
- Avinza: Subjects were prescribed Avinza at a QD (once daily) dose determined by the investigator and in adherence to the current Avinza prescribing information. Subjects were titrated on Avinza for up to one month and evaluated approximately 3 months at monthly visits once a stable dose was achieved. Avinza dosing was adjustable according to routine clinical practice, in order to achieve a balance of analgesia and opioid side effects. Avinza dose could not exceed 1600mg/day.
Period: Enrollment
Arm/Group | Avinza
Started | 1570 (Number of patients with evidence of prescription card receipt)
Completed | 1487 (Number of patients with evidence of study drug receipt)
Not Completed | 83
Not completed — Did not receive study drug | 83
Period: Treatment
Arm/Group | Avinza
Started | 1487
Completed | 561
Not Completed | 926

BASELINE CHARACTERISTICS:
Arm/Group | Avinza
Number analyzed (Participants) | 1487
Age Continuous [Mean (Standard Deviation); unit: years] | 52.7 (13.62)
Sex/Gender, Customized [Number; unit: participants]
  Female | 839
  Male | 630
  Missing | 18
Risk level for opioid misuse or abuse [Number; unit: participants] — Investigator determined classification of potential risk based on assessment of urine drug tests and patient history and questionnaires
  participants
    Low | 694
    Moderate | 767
    High | 19
    Missing | 7

OUTCOME MEASURES:

1. Primary Outcome: Difference From Baseline (Week 0) in the Average Pain Score at Visit 3 (Week 6)
Description: Average pain intensity over last 24 hours rated by the subject using an 11 point numeric rating scale (ranging from 0=no pain to 10=worst pain) at Visit 3
Time Frame: Baseline (Week 0) to Visit 3 (Week 6)
Population: Number of subjects with pain scores recorded at Baseline (Week 0) and Visit 3 (Week 6)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Avinza
Number analyzed (Participants) | 755
units on scale | -1.6 (2.27)

2. Primary Outcome: Difference From Baseline (Week 0) in the Average Pain Score at Visit 4 (Week 10)
Description: Average pain intensity over last 24 hours rated by the subject using an 11 point numeric rating scale (ranging from 0=no pain to 10=worst pain) at Visit 4
Time Frame: Baseline (Week 0) to Visit 4 (Week 10)
Population: Number of subjects with pain scores at Baseline (Week 0) and Visit 4 (Week 10)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Avinza
Number analyzed (Participants) | 622
units on scale | -1.7 (2.24)

3. Primary Outcome: Difference From Baseline (Week 0) in the Average Pain Score at Visit 5 (Week 14 / End of Study)
Description: Average pain intensity over last 24 hours rated by the subject using an 11 point numeric rating scale (ranging from 0=no pain to 10=worst pain) at Visit 5 / End of Study
Time Frame: Baseline (Week 0) to Visit 5 (Week 14 / End of Study)
Population: Number of subjects with pain scores at Baseline (Week 0) and Visit 5 (Week 14 / End of Study)
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Avinza
Number analyzed (Participants) | 1105
units on scale | -1.1 (2.31)

4. Primary Outcome: Number of Subjects With Treatment Emergent Adverse Events
Description: Adverse events that occur or worsen after the first dose of Avinza
Time Frame: Up to 4 months
Measure: Number; unit: participants
Arm/Group | Avinza
Number analyzed (Participants) | 1487
participants | 707

5. Primary Outcome: Number of Subjects at Each Level of Risk for Opioid Misuse or Abuse at Visit 3 (Week 6)
Description: Risk level was determined by the investigator using the subject's SOAPP-R (Screener and Opioid Assessment for Patients with Pain® - Revised Questionnaire) score, reports/ evidence of aberrant behavior and clinical judgment. Low Risk: SOAPP-R score <= 9 and no signals of aberrant behavior; Moderate Risk: SOAPP-R score <= 9 with positive signals of aberrant behavior OR SOAPP-R score = 10-21 with or without positive signals of aberrant behavior OR SOAPP-R score >= 22; High Risk: SOAPP-R score >= 22 with positive signals of aberrant behavior.
Time Frame: Visit 3 (Week 6)
Population: Number of subjects with risk level assessment at Visit 3 (Week 6)
Measure: Number; unit: participants
Arm/Group | Avinza
Number analyzed (Participants) | 769
participants
  Low risk | 433
  Moderate risk | 325
  High risk | 8
  Missing | 3

6. Primary Outcome: Number of Subjects at Each Level of Risk for Opioid Misuse or Abuse at Visit 4 (Week 10)
Description: Risk level was determined by the investigator using the subject's SOAPP-R score, reports/ evidence of aberrant behavior and clinical judgment. Low Risk: SOAPP-R score <= 9 and no signals of aberrant behavior; Moderate Risk: SOAPP-R score <= 9 with positive signals of aberrant behavior OR SOAPP-R score = 10-21 with or without positive signals of aberrant behavior OR SOAPP-R score >= 22; High Risk: SOAPP-R score >= 22 with positive signals of aberrant behavior.
Time Frame: Visit 4 (Week 10)
Population: Number of subjects with risk level assessment at Visit 4 (Week 10)
Measure: Number; unit: participants
Arm/Group | Avinza
Number analyzed (Participants) | 633
participants
  Low risk | 355
  Moderate risk | 267
  High risk | 7
  Missing | 4

7. Secondary Outcome: Number of Cases in Which Investigators Were Satisfied or Very Satisfied With the Utility of the Risk Minimization Program in This Study.
Description: After each subject completed participation in the study, investigators reported satisfaction with the utility of the risk minimization program in handling each subject's particular case. The risk minimization program is a set of tools used to assist clinicians in responsibly managing pain patients prescribed Avinza. The tools include SOAPP-R, treatment agreement, urine drug test, pill counts, PPAFT (Pain Patient Follow-up Tool), Investigator Assessment and Plan and prescription card data. These tools were used at each visit to assess subject risk and to aid in the management of subject's pain.
Time Frame: Up to 4 months
Population: Number of subjects with risk level assessment at Visit 4 (Week 10)
Measure: Number; unit: cases
Arm/Group | Avinza
Number analyzed (Participants) | 1487
cases
  Satisfied / Very Satisfied | 1010
  Neutral | 278
  Dissatisfied / Very dissatisfied | 56
  Missing | 143

8. Secondary Outcome: Number of Investigators Who Reported Continued Use of One or More Risk Minimization Tools Within 3 Months Post Study Completion.
Description: The risk minimization tools include SOAPP-R, treatment agreement, urine drug test, pill counts, PPAFT, Investigator Assessment and Plan and prescription card information.
Time Frame: 3 months post study
Population: Number of investigators providing 3-month post study survey response (n=219); surveys were completed one per investigator.
Measure: Number; unit: investigators
Arm/Group | Avinza
Number analyzed (Participants) | 219
investigators
  Use of at least one tool | 206
  Use of no tools | 13

9. Secondary Outcome: Number of Investigators Who Reported Continued Use of One or More Risk Minimization Tools Within 3 to 6 Months Post Study Completion.
Description: as for outcome 8
Time Frame: 6 months post study
Population: Number of investigators providing 6-month post study survey response (n=169); surveys were completed one per investigator.
Measure: Number; unit: investigators
Arm/Group | Avinza
Number analyzed (Participants) | 169
investigators
  Use of at least one tool | 156
  Use of no tools | 13

ADVERSE EVENTS:
Arm/Group | Avinza
Serious Adverse Events (participants affected / at risk) | 60/1487
Other Adverse Events (participants affected / at risk) | 394/1487
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avinza (N=1487)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 4 (4)
Myocardial infarction (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Accidential death (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Drug withdrawal syndrome (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Cellulitis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Respiratory rate decreased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3)
Syncope (Nervous system disorders) | 2 (2)
Complicated migraine (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 5 (5)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Shock (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avinza (N=1487)
Constipation (Gastrointestinal disorders) | 203 (218)
Nausea (Gastrointestinal disorders) | 162 (170)
Vomiting (Gastrointestinal disorders) | 78 (80)
Somnolence (Nervous system disorders) | 79 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results may only be published through Sponsor.